CLINICAL TRIAL: NCT04197232
Title: Study on the Safety for the Newborn of the Use of Biologics During Pregnancy
Brief Title: Study on the Safety for the Newborn of the Use of Biologics During Pregnancy by Mothers Affected by Autoimmune Diseases
Acronym: BIOGN1
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rosanna Rovelli, Principal Investigator, IRCCS San Raffaele
Other Study IDs: BIOGN1
Record Dates: First submitted 2019-11-27; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Suspected Damage to Fetus From Biologic Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed: The modality of study is a cohort study that evaluates the performance of children exposed to biologic agents during pregnancy compared to the performance of children born at the same gestational age not exposed to biologic agents.
- not exposed: The modality of study is a cohort study that evaluates the performance of children exposed to biologic agents during pregnancy compared to the performance of children born at the same gestational age not exposed to biologic agents.
  Interventions: Other: clinical evaluation

INTERVENTIONS:
Other: clinical evaluation — - In children: general clinical evaluation, birth weight, APGAR, ECG, admission to ICU, hospital admissions in perinatal age, presence of malformations; complete blood count, inflammatory index, complement, antibiotic treatment, brain ultra-sound, presence of infection, presence of sepsis, presence of necrotizing enterocolitis, growth curve, presence of recurrent infections, developmental milestones, response to vaccines, admission to hospital in the first year of life.
  Groups: not exposed

SUMMARY:
The goal of the study is to evaluate the effects on the offspring and therefore the safety of using biologic agents during pregnancy and their eventual consequences on children. The effects considered are divided into peri-partum and more long-term effects. Demonstration of safety in children born from mothers who received biologics during pregnancy will pave the way of their use in other women affected by autoimmune diseases unresponsive to standard treatment.

DETAILED DESCRIPTION:
Biologic agents are a group of genetically engineered drugs that target the immune system and have gained a lot of popularity in recent years. They act by interfering with cytokine function or production, inhibiting the "second signal" required for T-cell activation or by depleting B-cells. They are used for the treatment of a wide variety of diseases including Rheumatoid Arthritis, Psoriatic Arthritis, Systemic Lupus Erythematosus (SLE), some types of vasculitis and many more. Many of these pathologies occur in young women during child-bearing years and so it is important for these drugs to not only be safe to use for the patient but also during pregnancy for fetus and child. Many studies are conducted on their safety for the patients but few studies are present on the safety of use during pregnancy. There are even fewer studies that follow up for long term effects on the children outside of the perinatal period.

The goal of the study is to evaluate the effects on the offspring and therefore the safety of using biologic agents during pregnancy and their eventual consequences on children. The effects considered are divided into peri-partum and more long-term effects. Demonstration of safety in children born from mothers who received biologics during pregnancy will pave the way of their use in other women affected by autoimmune diseases unresponsive to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* children born from mothers treated with biologic agents

Exclusion Criteria:

-

Ages: 1 Day to 12 Years | Sex: All
Age Groups: Child
Study Population: children born from mothers treated with biologic agents during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety on fetus of biologic agents used during pregnancy | 8 years
  Evaluation of increased incidence of preterm births (measured by gestational age at birth (gestational weeks)
Safety on fetus of biologic agents used during pregnancy - fetal development | 8 years
  Evaluation of normal intrauterine development (measured by presence of Intra-Uterine Growth Restriction, presence of malformations (number#), birth weight (grams), length (cm), head circumference (cm))
Safety on fetus of biologic agents used during pregnancy - adequate growth for GA | 8 years
  Evaluation of normal intrauterine development - birth weight (grams), length (cm), head circumference (cm))
Safety on fetus of biologic agents used during pregnancy - perinatal complications | 8 years
  Evaluation of increased rate of perinatal complications (measured by: admission to ICU (number#), hospital admissions in perinatal) (number#)
Safety on fetus of biologic agents used during pregnancy - neurological development | 8 years
  Evaluation of developmental milestones (age in months of acquisition of head control, sitting position, crawling and standing position)
Safety on fetus of biologic agents used during pregnancy - immunological evaluation | 8 years
  Evaluation of immunological status (complete blood count (absolute counts od WBC, Lymphocytes and Neutrophilis), presence of infection (number #), response to vaccines (presence/absence)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS ospedale san raffaele, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No